CLINICAL TRIAL: NCT00301925
Title: Trial of Accelerated Adjuvant Chemotherapy With Capecitabine in Early Breast Cancer (TACT2)
Brief Title: Combination Chemotherapy in Treating Patients With Early Stage Breast Cancer That Has Been Removed By Surgery
Acronym: TACT2
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Purpose: Treatment
Other Study IDs: CDR0000463447; ICR-TACT2; EU-205114; EUDRACT-2004-000066-13; MREC-04/MRE00/88; ISRCTN68068041
Record Dates: First submitted 2006-03-09; First posted 2006-03-13 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — pegfilgrastim; Capecitabine; Cyclophosphamide; Epirubicin; Fluorouracil; Methotrexate; Chemotherapy, Adjuvant

ARMS (4):
- Epi-CMF (Active Comparator)
  Interventions: Drug: cyclophosphamide; Drug: epirubicin hydrochloride; Drug: fluorouracil; Drug: methotrexate; Procedure: adjuvant therapy
- Accelerated Epi-CMF (Experimental)
  Interventions: Biological: pegfilgrastim; Drug: cyclophosphamide; Drug: epirubicin hydrochloride; Drug: fluorouracil; Drug: methotrexate; Procedure: adjuvant therapy
- Epi-Capecitabine (Experimental)
  Interventions: Drug: capecitabine; Drug: epirubicin hydrochloride; Procedure: adjuvant therapy
- Accelerated Epi-Capecitabine (Experimental)
  Interventions: Biological: pegfilgrastim; Drug: capecitabine; Drug: epirubicin hydrochloride; Procedure: adjuvant therapy

INTERVENTIONS:
Biological: pegfilgrastim
  Arms: Accelerated Epi-CMF; Accelerated Epi-Capecitabine
Drug: capecitabine
  Arms: Accelerated Epi-Capecitabine; Epi-Capecitabine
Drug: cyclophosphamide
  Arms: Accelerated Epi-CMF; Epi-CMF
Drug: epirubicin hydrochloride
Drug: fluorouracil
  Arms: Accelerated Epi-CMF; Epi-CMF
Drug: methotrexate
  Arms: Accelerated Epi-CMF; Epi-CMF
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Giving combination chemotherapy after surgery may kill any remaining tumor cells. It is not yet known which combination chemotherapy regimen is more effective in treating early stage breast cancer that has been removed by surgery.

PURPOSE: This randomized phase III trial is studying four different combination chemotherapy regimens to compare how well they work in treating patients with early stage breast cancer that has been removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the disease-free survival (DFS) of patients with completely resected early stage breast cancer receiving 1 of 2 different schedules of adjuvant chemotherapy comprising epirubicin, cyclophosphamide, methotrexate, and fluorouracil versus 1 of 2 different schedules of adjuvant chemotherapy comprising epirubicin and capecitabine.

Secondary

* Compare overall survival (OS) and distant disease-free survival (DFS).
* Compare the tolerability (including serious adverse events [SAE], dose-intensity, and toxicity) of these regimens.
* Determine the detailed toxicity of these regimens.
* Determine the quality of life of a subset of these patients.

OUTLINE: This is a multi-center, randomized study. Patients are stratified according to participating center, nodal status (N0 vs N1-3 vs N≥ 4), age (≤ 50 years vs > 50 years), and estrogen receptor (ER) status (negative vs positive). Patients are randomized to 1 of 4 treatment arms.

* Arm I: Patients receive epirubicin on day 1. Treatment repeats every 3 weeks for 4 courses. Patients then receive cyclophosphamide orally once daily on days 1-14 or IV on days 1 and 8 and methotrexate and fluorouracil on days 1 and 8. Treatment repeats every 28 days for 4 courses.
* Arm II: Patients receive epirubicin on day 1 and pegfilgrastim on day 2. Treatment repeats every 2 weeks for 4 courses. Patients then receive cyclophosphamide, methotrexate and fluorouracil as in arm I.
* Arm III: Patients receive epirubicin as in arm I. Patients then receive oral capecitabine twice daily on days 1-14. Treatment with capecitabine repeats every 3 weeks for 4 courses.
* Arm IV: Patients receive epirubicin and pegfilgrastim as in arm II. Patients then receive capecitabine as in arm III.

In all arms, treatment continues in the absence of unacceptable toxicity.

Beginning 3-6 months later, all patients may undergo radiotherapy at the discretion of the principal investigator. Patients with ER- and/or progesterone receptor-positive disease then receive tamoxifen citrate or an aromatase inhibitor for up to 5 years.

Quality of life is assessed in a cohort of 1,000 patients in week 6, week 8 or 12, and week 20 or 24 during treatment and then at 12 and 24 months after randomization.

After completion of study therapy, patients are followed every 6 months for 2 years and then annually for at least 10 years.

Peer Reviewed and Funded or Endorsed by Cancer Research UK.

PROJECTED ACCRUAL: A total of 4,400 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histological diagnosis of invasive breast carcinoma

  * Cytological proof of malignancy alone is not sufficient
  * Early stage disease (T0-3, N0-2, M0) without clinical suspicion or evidence of distant metastases on routine staging
  * No locally advanced breast cancer (T4 and/or N3 disease)
* Completely resected disease by breast-conserving surgery with axillary node clearance or modified radical mastectomy within the past 4-8 weeks

  * Negative surgical margins required, unless either of the following are true:

    * Deep surgical margins after full thickness resection
    * Noninvasive cancer at surgical margins for which a mastectomy is planned after completion of study chemotherapy
  * No contraindication for or refusal of postoperative radiotherapy in patients who underwent prior breast-conserving surgery
* Definite indication for adjuvant chemotherapy
* No prior or current invasive breast cancer or bilateral breast cancer

  * Prior surgically-treated ductal carcinoma in situ or lobular carcinoma in situ allowed
* Hormone receptor status:

  * Estrogen receptor- and/or progesterone receptor-positive or -negative tumor

PATIENT CHARACTERISTICS:

* Sex: male or female
* Menopausal status: premenopausal or postmenopausal
* No previous malignancy except basal cell carcinoma, carcinoma in situ of the cervix, or any cancer from which the patient has been disease-free for 10 years and for which treatment consisted solely of resection
* ECOG status 0 or 1
* Hemoglobin > 9 g/dL
* WBC > 3,000/mm³
* Platelet count > 10,000/mm³
* Bilirubin normal (unless due to known Gilbert's disease)
* AST and ALT ≤ 1.5 times upper limit of normal (ULN)
* Albumin normal
* Creatinine ≤ 1.5 times ULN
* Creatinine clearance > 50 mL/min
* No active, uncontrolled infection
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No concurrent medical, psychiatric, or geographic problems that might prevent completion of treatment or follow-up
* Available for a minimum of 5 years' follow-up
* No known serious viral infection such as active hepatitis B, hepatitis C, or HIV
* No significant cardiac disease, such as impaired left ventricular function or active angina requiring regular anti-anginal medication and/or resulting in restricted physical activity
* No history of significant renal impairment or disease

PRIOR CONCURRENT THERAPY:

* No simultaneous participation in the active intervention phase of another treatment trial
* Not being approached or recruited for another trial within 2 months of study entry
* No previous chemotherapy, hormonal therapy or radiotherapy for the treatment of pre-invasive or invasive cancer except for either of the following:

  * Previous radiotherapy for basal cell carcinoma
  * Previous preoperative endocrine therapy, provided there was no evidence of progression during this therapy, it lasted for less than 6 weeks in duration, and it was stopped at least one month prior to trial entry
* Concurrent luteinizing hormone-releasing hormone analog therapy allowed for premenopausal patients
* More than 4 weeks since prior hormone replacement therapy (HRT) or pre-operative endocrine therapy
* No prior breast conserving surgery if there is a contradiction for or refusal of postoperative radiotherapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4400 (Estimated)
Dates: Start 2005-12-16 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) at 5 years

SECONDARY OUTCOMES:
Overall survival at 5 years
Distant DFS at 5 years
Tolerability (including serious adverse events, dose-intensity, and toxicity)
Detailed toxicity
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: David Cameron, MD, Study Chair — National Cancer Research Network
Locations (152):
- United Kingdom (152):
  - William Harvey Hospital, Ashford-Kent, England
  - Wansbeck General Hospital, Ashington, England
  - Tameside General Hospital, Ashton-under-Lyne, England
  - North Devon District Hospital, Barnstaple, England
  - Furness General Hospital, Barrow in Furness, England
  - Basildon University Hospital, Basildon, England
  - Basingstoke and North Hampshire NHS Foundation Trust, Basingstoke, England
  - Queen Elizabeth Hospital at University Hospital of Birmingham NHS Trust, Birmingham, England
  - City Hospital - Birmingham, Birmingham, England
  - Birmingham Heartlands Hospital, Birmingham, England
  - Royal Blackburn Hospital, Blackburn, England
  - Blackpool Victoria Hospital, Blackpool, England
  - Royal Bolton Hospital, Bolton, Lancashire, England
  - Bradford Royal Infirmary, Bradford, England
  - Sussex Cancer Centre at Royal Sussex County Hospital, Brighton, England
  - Bristol Haematology and Oncology Centre, Bristol, England
  - Broomfield Hospital, Broomefield, England
  - Burnley General Hospital, Burnley, England
  - Queen's Hospital, Burton-on-Trent, England
  - West Suffolk Hospital, Bury St Edmunds, England
  - Addenbrooke's Hospital, Cambridge, England
  - Kent and Canterbury Hospital, Canterbury, England
  - Cheltenham General Hospital, Cheltenham, England
  - Halton Hospital, Cheshire, England
  - Chesterfield Royal Hospital, Chesterfield, England
  - Saint Richards Hospital, Chichester, England
  - Essex County Hospital, Colchester, England
  - Walsgrave Hospital, Coventry, England
  - Darent Valley Hospital, Dartford Kent, England
  - Derbyshire Royal Infirmary, Derby, England
  - Dewsbury and District Hospital, Dewsbury, England
  - Doncaster Royal Infirmary, Doncaster, England
  - Russells Hall Hospital, Dudley, England
  - University Hospital of North Durham, Durham, England
  - Eastbourne District General Hospital, Eastbourne, England
  - Royal Devon and Exeter Hospital, Exeter, England
  - Queen Elizabeth Hospital, Gateshead, England
  - Gloucestershire Royal Hospital, Gloucester, England
  - Diana Princess of Wales Hospital, Grimsby, England
  - St. Luke's Cancer Centre at Royal Surrey County Hospital, Guildford, England
  - UCL Cancer Institute, Hampstead, London, England
  - Hereford Hospitals NHS Trust, Hereford, England
  - Wycombe General Hospital, High Wycombe, England
  - Huddersfield Royal Infirmary, Huddersfield, West Yorks, England
  - Princess Royal Hospital at Hull and East Yorkshire NHS Trust, Hull, England
  - King George Hospital, Ilford, Essex, England
  - Ipswich Hospital, Ipswich, England
  - West Middlesex University Hospital, Isleworth, England
  - Airedale General Hospital, Keighley, England
  - Kettering General Hosptial, Kettering, Northants, England
  - Kidderminster Hospital, Kidderminster Worcestershire, England
  - Queen Elizabeth Hospital, Kings Lynn, England
  - Royal Albert Edward Infirmary, Lancanshire, England
  - Royal Lancaster Infirmary, Lancaster, England
  - Cookridge Hospital, Leeds, England
  - National Cancer Research Network, Leeds, England
  - Cancer Research UK Clinical Centre at St. James's University Hospital, Leeds, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Royal Liverpool University Hospital, Liverpool, England
  - Aintree University Hospital, Liverpool, England
  - Barts and the London School of Medicine, London, England
  - Whittington Hospital, London, England
  - University College Hospital, London, England
  - Guy's Hospital, London, England
  - King's College Hospital, London, England
  - St. George's Hospital, London, England
  - St. Mary's Hospital, London, England
  - Charing Cross Hospital, London, England
  - Macclesfield District General Hospital, Macclesfield, England
  - Maidstone Hospital, Maidstone, England
  - Christie Hospital, Manchester, England
  - Withington Hospital, Manchester, England
  - North Manchester General Hospital - Penine Actute Hospitals Trust, Manchester, England
  - Queen Elizabeth The Queen Mother Hospital, Margate, England
  - Clatterbridge Centre for Oncology, Merseyside, England
  - James Cook University Hospital, Middlesbrough, England
  - Northern Centre for Cancer Treatment at Newcastle General Hospital, Newcastle upon Tyne, England
  - St. Mary's Hospital, Newport, England
  - James Paget Hospital, Norfolk, England
  - North Tyneside Hospital, North Shields, England
  - Friarage Hospital, North Yorks, England
  - Northampton General Hospital NHS Trust, Northampton, England
  - Norfolk and Norwich University Hospital, Norwich, England
  - Nottingham City Hospital NHS Trust, Nottingham, England
  - King's Mills Hospital, Nottinghamshire, England
  - George Eliot Hospital, Nuneaton, England
  - Royal Oldham Hospital, Oldham, England
  - Radcliffe Infirmary NHS Trust, Oxford, England
  - Churchill Hospital, Oxford, England
  - Peterborough Hospitals Trust, Peterborough, England
  - Pontefract General Infirmary, Pontefract West Yorkshire, England
  - Whiston Hospital, Prescot Merseyside, England
  - Royal Preston Hospital, Preston, England
  - Alexandra Healthcare NHS, Redditch, Worcestershire, England
  - Oldchurch Hospital, Romford, England
  - Conquest Hospital, Saint Leonards-on-Sea, England
  - Salisbury District Hospital, Salisbury, England
  - Scunthorpe General Hospital, Scunthorpe, England
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - Royal Shrewsbury Hospital, Shrewsbury, England
  - Solihull Hospital, Solihull, England
  - Southampton General Hospital, Southampton, England
  - Southport and Formby District General Hospital, Southport, England
  - Stepping Hill Hospital, Stockport, England
  - University Hospital of North Staffordshire, Stoke-on-Trent, England
  - Sunderland Royal Hospital, Sunderland, England
  - Great Western Hospital, Swindon, England
  - Taunton and Somerset Hospital, Taunton, England
  - Torbay Hospital, Torquay, England
  - Royal Cornwall Hospital, Truro, Cornwall, England
  - Walsall Manor Hospital, Walsall, England
  - Warrington Hospital NHS Trust, Warrington, England
  - South Warwickshire Hospital, Warwick, Warwickshire, England
  - Sandwell General Hospital, West Bromwich, England
  - Southend University Hospital NHS Foundation Trust, Westcliff-on-Sea, England
  - Weston General Hospital, Weston-super-Mare, England
  - Royal Hampshire County Hospital, Winchester, England
  - New Cross Hospital, Wolverhampton, England
  - Worcester Royal Hospital, Worcester, England
  - Yeovil District Hospital, Yeovil - Somerset, England
  - Belfast City Hospital Trust Incorporating Belvoir Park Hospital, Belfast, Northern Ireland
  - Centre for Cancer Research and Cell Biology at Queen's University Belfast, Belfast, Northern Ireland
  - Altnagelvin Area Hospital, Londonderry, Northern Ireland
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Ayr Hospital, Ayr, Scotland
  - Dumfries & Galloway Royal Infirmary, Dumfries, Scotland
  - Ninewells Hospital, Dundee, Scotland
  - Queen Margaret Hospital - Dunfermline, Dunfermline, Scotland
  - Hairmyres Hospital, East Kilbride, Scotland
  - Edinburgh Cancer Centre at Western General Hospital, Edinburgh, Scotland
  - Dr Gray's Hospital, Elgin, Scotland
  - Falkirk & District Royal Infirmary, Falkirk, Scotland
  - Beatson West of Scotland Cancer Centre, Glasgow, Scotland
  - Royal Infirmary - Castle, Glasgow, Scotland
  - Inverclyde Royal Hospital, Greenock, Scotland
  - Raigmore Hospital, Inverness, Scotland
  - Crosshouse Hospital, Kilmarnock, Scotland
  - St. John's Hospital, Livingston, Scotland
  - Scarborough General Hospital, Scarborough, Scotland
  - Pinderfields General Hospital, Wakefield, Scotland
  - Wishaw General Hospital, Wishaw, Scotland
  - Bronglais District General Hospital, Aberystwyth, Wales
  - Ysbyty Gwynedd, Bangor, Wales
  - Princess of Wales Hospital, Bridgend, Wales
  - Velindre Cancer Center at Velindre Hospital, Cardiff, Wales
  - Withybush General Hospital, Haverfordwest, Wales
  - Royal Glamorgan Hospital, Lhantrisant, Wales
  - Prince Charles Hospital, Mid Glamorgan, Wales
  - Royal Gwent Hospital, Newport Gwent, Wales
  - Glan Clwyd Hospital, Rhyl, Denbighshire, Wales
  - Wrexham Maelor Hospital, Wrexham, Wales
  - Barnet General Hospital, Barnet, Hertfordshire

REFERENCES:
- [Derived] Velikova G, Morden JP, Haviland JS, Emery C, Barrett-Lee P, Earl H, Bloomfield D, Brunt AM, Canney P, Coleman R, Verrill M, Wardley A, Bertelli G, Ellis P, Stein R, Bliss JM, Cameron D; TACT2 Trial Management Group. Accelerated versus standard epirubicin followed by cyclophosphamide, methotrexate, and fluorouracil or capecitabine as adjuvant therapy for breast cancer (UK TACT2; CRUK/05/19): quality of life results from a multicentre, phase 3, open-label, randomised, controlled trial. Lancet Oncol. 2023 Dec;24(12):1359-1374. doi: 10.1016/S1470-2045(23)00460-6. Epub 2023 Nov 2. PMID 37926100
- [Derived] Hoon SN, Lau PK, White AM, Bulsara MK, Banks PD, Redfern AD. Capecitabine for hormone receptor-positive versus hormone receptor-negative breast cancer. Cochrane Database Syst Rev. 2021 May 26;5(5):CD011220. doi: 10.1002/14651858.CD011220.pub2. PMID 34037241
- [Derived] Cameron D, Morden JP, Canney P, Velikova G, Coleman R, Bartlett J, Agrawal R, Banerji J, Bertelli G, Bloomfield D, Brunt AM, Earl H, Ellis P, Gaunt C, Gillman A, Hearfield N, Laing R, Murray N, Couper N, Stein RC, Verrill M, Wardley A, Barrett-Lee P, Bliss JM; TACT2 Investigators. Accelerated versus standard epirubicin followed by cyclophosphamide, methotrexate, and fluorouracil or capecitabine as adjuvant therapy for breast cancer in the randomised UK TACT2 trial (CRUK/05/19): a multicentre, phase 3, open-label, randomised, controlled trial. Lancet Oncol. 2017 Jul;18(7):929-945. doi: 10.1016/S1470-2045(17)30404-7. Epub 2017 Jun 7. PMID 28600210